CLINICAL TRIAL: NCT07398313
Title: Effectiveness Of Prehabilitation On Pelvic Floor Weakness, Functional Performance And Recovery Efficiency Among Post-Surgical Cervical Cancer Women
Brief Title: Effect of Prehabilitation on Recovery Outcomes in Post-Surgical Cervical Cancer Women
Acronym: PROP-CC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saveetha University (Other)
Responsible Party: Principal Investigator, Akshya Sam, Principal Investigator, Post Graduate Student , Department of Community, Geriatric and Palliative care Physiotherapy, SIMATS college of Physiotherapy, SIMATS., Saveetha University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 063/05/2025/ISRB/PGSR/SCPT
Record Dates: First submitted 2026-01-14; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Cervical Adenocarcinoma; Hysterectomy; Cervical Cancer
Keywords: Prehabilitation; Cervical Cancer; Pelvic floor; Functional performance; Recovery Efficiency; hysterectomy
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Congresses as Topic

STUDY DESIGN:
Intervention Model Description: This randomized controlled,evaluated the effectiveness of prehabilitation on pelvic floor weakness, functional performance and recovery efficiency in post-surgical cervical cancer women. The study was conducted in the inpatient and outpatient departments of a hospital. Women aged 40-60 years with early-stage cervical cancer scheduled for radical hysterectomy and a Karnofsky Performance Scale score of 50-70 were eligible. Of 46 patients screened, 39 were randomized using the lottery method into a prehabilitation group (n = 19) or control group (n = 20). Baseline assessments included Brink score, Karnofsky Performance Scale and hospital stay. The prehabilitation group received four weeks of structured aerobic, resistance and pelvic floor exercises, while controls received conventional care. Both groups underwent identical postoperative rehabilitation. Post-test assessment followed two weeks post-surgery. Non-parametric analysis was performed (p < 0.05). No adverse events were reported.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prehabilitation Group (Experimental): The program consisted of three supervised sessions per day, each lasting 20 minutes, amounting to 60 minutes of daily exercise. Aerobic training included walking, cycling or treadmill exercises based on individual tolerance, pelvic floor muscle training was performed as two sets of ten repetitions focusing on proper activation and endurance and resistance training targeted upper and lower limb muscle groups using resistance bands, dumbbells, weight cuffs and a Swiss ball. Exercise intensity and progression were individualized according to each participant's functional capacity.
  Interventions: Behavioral: Structured Prehabilitation Protocol
- Control Group (Active Comparator): The control group received conventional preoperative care for the same duration, which included free exercises, breathing exercises and walking, without structured resistance or pelvic floor-specific training.
  Interventions: Behavioral: Conventional

INTERVENTIONS:
Behavioral: Structured Prehabilitation Protocol — The prehabilitation intervention in this study is distinguished by its multimodal, time-bound and individualized design delivered during the preoperative window. Unlike conventional preoperative care, the program integrated aerobic conditioning, progressive resistance training and targeted pelvic floor muscle training with a structured 4-week protocol, providing 60 minutes of supervised daily exercise. Pelvic floor training emphasized correct muscle activation, endurance and coordination using standardized repetitions, while resistance exercises targeted both upper and lower limb muscle groups with graded external resistance. Exercise intensity and progression were individualized based on functional capacity, ensuring feasibility for women with moderate functional limitation. Both study groups received identical postoperative rehabilitation, allowing the isolated effect of prehabilitation on recovery outcomes,differentiating this intervention from other perioperative studies.
  Arms: Prehabilitation Group
Behavioral: Conventional — The control group received conventional preoperative care for the same duration, which included free exercises, breathing exercises and walking, without structured resistance or pelvic floor-specific training.
  Arms: Control Group

SUMMARY:
This randomized controlled trial was conducted among patients diagnosed with cervical cancer and scheduled to undergo radical hysterectomy. A total of 34 participants were recruited using a simple random sampling technique after obtaining approval from the Institutional Ethics Committee. Participants were screened based on predefined selection criteria to ensure safety, reliability of outcome measures and avoidance of confounding medical conditions. Eligible patients were informed in detail about the study, and written informed consent was obtained prior to enrollment.

Participants were randomly allocated into two equal groups (n = 17 each) using the lottery method, with allocation concealment maintained to minimize selection bias. Baseline assessments were carried out four weeks prior to surgery and included evaluation of pelvic floor muscle strength using the Brink score, functional status using the Karnofsky Performance Scale and anticipated duration of hospital stay as an indicator of recovery efficiency.

The intervention group underwent a structured prehabilitation exercise program for four weeks before surgery, consisting of three supervised daily sessions totaling 60 minutes. The program included aerobic training, targeted pelvic floor muscle strengthening and upper and lower limb resistance training, with exercise intensity and progression individualized according to the participant's functional capacity. The control group received a generalized standard exercise protocol comprising free exercises, breathing exercises and walking, delivered with similar session duration but without structured resistance or pelvic floor-specific training.

Postoperatively, both groups received a standardized rehabilitation program for two weeks, including breathing exercises, pelvic floor strengthening and core stabilization exercises to promote early mobilization and prevent complications. Post-intervention assessments were conducted after two weeks to evaluate the effectiveness of the intervention. The study utilized basic exercise and assessment equipment, including resistance bands, weight cuffs, dumbbells, a Swiss ball, a couch and a stopwatch.

DETAILED DESCRIPTION:
Subjects: Patients with cervical cancer undergoing radical hysterectomy. Sampling technique: Simple random sampling technique Sample size: 34 Selection criteria: The selection criteria for the present study were carefully formulated to ensure the inclusion of participants who could safely undergo the intervention and provide reliable outcome data, while excluding individuals with conditions that could confound the results or pose medical risks. The criteria were applied uniformly during participant screening prior to enrollment.

Study procedure: After obtaining approval from the Institutional Ethics Committee, the study was conducted as a randomized controlled trial among patients diagnosed with cervical cancer and scheduled to undergo radical hysterectomy. The study setting included the inpatient and outpatient departments. Potential participants were screened by the investigator based on the predefined inclusion and exclusion criteria. Eligible participants were approached individually and a detailed explanation of the study objectives, procedures, potential benefits and possible risks was provided in a language understandable to them. Adequate time was given for clarification of doubts following which written informed consent was obtained prior to enrolment in the study.

A total of 34 participants who satisfied the selection criteria were included. Simple random sampling was adopted for participant selection and random allocation into two groups was carried out using the lottery method to ensure unbiased group assignment. The participants were equally divided into two groups, the intervention group and the control group, with 17 participants in each group. Allocation concealment was maintained throughout the recruitment process to minimize selection bias.

Baseline assessments were conducted four weeks prior to the scheduled surgical procedure. Pre-test measurements included assessment of pelvic floor muscle strength using the Brink score, evaluation of overall functional status using the Karnofsky Performance Scale and assessment of recovery efficiency through the anticipated duration of hospital stay. All baseline assessments were performed before the commencement of the exercise intervention to ensure uniformity in data collection.

Participants allocated to the intervention group underwent a structured prehabilitation exercise program for a duration of four weeks prior to surgery. The prehabilitation protocol consisted of three supervised sessions per day, each lasting 20 minutes, amounting to a total of 60 minutes of exercise daily. The first session focused on aerobic training, which included activities such as walking, cycling and treadmill exercises based on the individual's choice, tolerance and fitness level. The second session emphasized pelvic floor muscle strengthening exercises, which were individualized and performed as two sets of ten repetitions to improve pelvic floor muscle activation and endurance. The third session consisted of resistance training exercises targeting both upper and lower limb muscle groups using appropriate equipment also performed as two sets of ten repetitions. Exercise intensity and progression were individualized based on the participant's functional capacity and clinical status.

Participants in the control group received a generalized standard exercise protocol for four weeks prior to surgery. This protocol included free exercises, breathing exercises and walking, delivered in three daily sessions similar in duration to the intervention group. However, no structured or targeted prehabilitation components such as resistance training or specific pelvic floor muscle strengthening were included in the control protocol.

Following surgery, participants in both groups underwent standardized postoperative rehabilitation for a period of two weeks. Postoperative rehabilitation included breathing exercises, pelvic floor strengthening exercises such as Kegel exercises and pelvic bridging and core strengthening exercises aimed at promoting early mobilization, improving functional recovery and preventing postoperative complications. The postoperative rehabilitation protocol was uniform for both groups to ensure comparability. Post-intervention assessments were conducted as per the study timeline after two weeks to evaluate the effectiveness of the intervention.

Materials Required: The materials required for the study included basic exercise and assessment equipment. For the intervention group, resistance bands, weight cuffs, dumbbells and a Swiss ball were used to perform aerobic, resistance and pelvic floor strengthening exercises. For outcome assessment, a couch and a stopwatch were used to facilitate standardized functional and pelvic floor muscle evaluations.

ELIGIBILITY:
Inclusion Criteria:

* Women aged between forty and sixty years
* Confirmed diagnosis of cervical cancer
* Preoperative diagnosis of early-stage cervical cancer
* Planned to undergo radical hysterectomy
* Karnofsky Performance Scale score between 50 and 70
* Ability to actively engage in pelvic floor and resistance training protocols
* Willingness to participate in the study
* Provision of written informed consent prior to inclusion

Exclusion Criteria:

* Diagnosis of locally advanced or metastatic cervical cancer
* Presence of cardiopulmonary comorbidities limiting exercise tolerance
* Active urinary tract infection at the time of assessment
* Cognitive impairments interfering with understanding or compliance with the intervention
* Any medical condition contraindicating participation in structured exercise programs

Ages: 40 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — female
Enrollment: 34 (Actual)
Dates: Start 2025-06-17 (Actual); Primary Completion 2025-10-07 (Actual); Study Completion 2025-11-22 (Actual)

PRIMARY OUTCOMES:
Pelvic floor muscle strength using the Brink score | baseline at four weeks prior surgery and post test assessment two week after surgery
  The Brink Score was used to evaluate pelvic floor muscle strength. The Brink score is a digital vaginal palpation scale used to assess pelvic floor muscle function by evaluating pressure (strength), duration (endurance), and vertical displacement (lift). With the patient in supine or crook-lying position, a gloved finger is inserted vaginally and the patient is instructed to contract the pelvic floor muscles. Each component is scored from 0 to 4, giving a total score of 0-12. Scores of 0-3 indicate severe weakness, 4-6 moderate weakness, 7-9 fair strength and 10-12 strong pelvic floor muscles.
Functional performance using the Karnofsky Performance Scale | baseline at four weeks prior surgery and post test assessment two week after surgery
  The Karnofsky Performance Scale is a standardized tool used to assess a patient's functional status and ability to perform daily activities, particularly in oncology and chronic illness care. KPS is widely used to evaluate disease severity, prognosis, treatment tolerance, and eligibility for therapies, and to monitor changes in functional capacity over time.
Recovery efficiency through hospital stay duration | baseline at four weeks prior surgery and post test assessment two week after surgery
  The duration of hospital stay was used as a measure of recovery efficiency. It was calculated as the number of days from the date of surgery to the date of hospital discharge, as documented in medical records. Shorter hospital stay was interpreted as improved recovery and functional readiness for discharge.

CONTACTS AND LOCATIONS:
Locations (1):
- SaveethaUniversity, Chennai, Tamil Nadu, India

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2025-05-09): https://cdn.clinicaltrials.gov/large-docs/13/NCT07398313/Prot_SAP_ICF_000.pdf